CLINICAL TRIAL: NCT03903302
Title: A Single Center, Randomised Study to Investigate Pharmacokinetics of CS1, Safety and Tolerability and in Obese, Borderline Hypertensive But Otherwise Healthy and Medicine Free Subjects After Administration of Single and Multiple Doses
Brief Title: Study Investigation Pharmacokinetics and Pharmacodynamics of CS1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cereno Scientific AB (Industry)
Responsible Party: Principal Investigator, Jan Erik Berglund, Principle Investigator, Cereno Scientific AB
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS1-001; 2017-002140-32 (EudraCT Number)
Record Dates: First submitted 2019-03-29; First posted 2019-04-04 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Thrombosis
Keywords: tissue-plasminogen activator (t-PA); plasminogen-activator inhibitor 1 (PAI-1); fibrinolysis; thrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Intervention Model Description: Safety, pharmacokinetics and pharmacodynamics of CS1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CS 1 I SAD (Active Comparator): Single dose pharmacokinetics of CS1 I
  Interventions: Drug: CS1-Sodium Valproate
- CS 1 II SAD (Active Comparator): Single dose pharmacokinetics of CS1 II
  Interventions: Drug: CS1-Sodium Valproate
- CS 1 III SAD (Active Comparator): Single dose pharmacokinetics of CS1 III
  Interventions: Drug: CS1-Sodium Valproate
- CS 1 II MAD (Active Comparator): Multiple dose pharmacokinetics of CS1 II
  Interventions: Drug: CS1-Sodium Valproate

INTERVENTIONS:
Drug: CS1-Sodium Valproate — Single and multiple dose evaluation of CS1

SUMMARY:
SAD study:

Eighteen subjects will be included in the SAD study (single dose) in 3 parallel arms, each with 6 subjects. The 3 arms will receive a single dose of one of the CS1 formulations I, II or III. The result of the pharmacokinetics analysis from the 6 first subjects is defined as SAD Pilot and will be used to evaluate the timing of PK sampling. Based on pharmacokinetic evaluations from all 18 subjects one of the formulations I (275 mg), II (276 mg) or III (276 mg) will be chosen to proceed into the MAD study. If none of the formulations show the desired PK properties the formulations may be re-dosed with a slightly different timing of the dose, i.e the IMP to be administered earlier or later during the evening.

MAD study:

Fifteen subjects will be included in a dose escalating study with 2 dose levels. The subjects will receive the lowest dose level (275 or 276 mg depending on the outcome of SAD) for the first 2 weeks before the dose is doubled (550 or 552 mg depending on the outcome of SAD) for the following 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study
2. Male and female subjects age ≥ 40 years, ≤ 75 years inclusive.
3. BMI 27- 35 kg/m2
4. PAI-1 levels minimum 15 kIE/L (applies only to the MAD study)
5. Acceptable medical history, physical findings, vital signs, ECG and laboratory values at the time of screening, as judged by the Investigator. Subjects with stable hypertension with one or more antihypertensive drugs can be accepted as acceptable medical history.
6. Male subjects who has not documented a vasectomy, must be willing to use condom from the date of dosing until three months after dosing of the IMP to prevent drug exposure of a partner and refrain from donating sperm and if they have a fertile partner, she must use contraceptive methods with a failure rate of < 1% to prevent pregnancy .
7. The females must be of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or post-menopausal defined as 12 months of amenorrhea (simultaneous determination of follicle stimulating hormone 25-140 IU/l and estradiol < 200 pmol/l is confirmatory) -

Exclusion Criteria:

Diagnosis and main eligibility criteria

Inclusion criteria:

1. Willing and able to give written informed consent for participation in the study
2. Male and female subjects age ≥ 40 years, ≤ 75 years inclusive.
3. BMI 27- 35 kg/m2
4. PAI-1 levels minimum 15 kIE/L (applies only to the MAD study)
5. Acceptable medical history, physical findings, vital signs, ECG and laboratory values at the time of screening, as judged by the Investigator. Subjects with stable hypertension with one or more antihypertensive drugs can be accepted as acceptable medical history.
6. Male subjects who has not documented a vasectomy, must be willing to use condom from the date of dosing until three months after dosing of the IMP to prevent drug exposure of a partner and refrain from donating sperm and if they have a fertile partner, she must use contraceptive methods with a failure rate of < 1% to prevent pregnancy .
7. The females must be of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or post-menopausal defined as 12 months of amenorrhea (simultaneous determination of follicle stimulating hormone 25-140 IU/l and estradiol < 200 pmol/l is confirmatory)

Exclusion criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. Subjects with active or chronic liver disease or personal or familiar history of drug related severe hepatic dysfunction.
3. Subjects with phorphyria.
4. Subjects with Systemic lupus erytematosus (SLE)
5. Subjects with TPK, APTT, INR levels which are significant outside the reference intervals as judged by the investigator.
6. History of severe bleeding disease or thrombotic disease.
7. Subjects on regular treatment with anticoagulant or antiplatelets drugs
8. Subjects with significant cardiac disease.
9. Subjects with significant pancreatic disease.
10. Subjects with gastrointestinal problems/ diseases e.g. inflammatory bowel disease and irritable bowel syndrome
11. Any clinically significant illness, medical/surgical procedure or trauma within four weeks of the first administration of IMP.
12. Any planned major surgery within the duration of the study.
13. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody and Human Immunodeficiency Virus (HIV).
14. After 10 minute supine rest at the time of screening, any vital signs values outside the following ranges:

    * Systolic blood pressure > 160 mm Hg
    * Diastolic blood pressure > 100 mm Hg
    * Heart rate < 40 or > 90 beats per minute
15. Prolonged QTcF (>450 ms), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG at the time of screening, as judged by the Investigator.
16. History of severe allergy/hypersensitivity or on-going allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to valproate acid or any other ingredient of the investigational medicinal product.
17. Administration of another new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical study that included drug treatment with less than three months between administration of last dose and first dose of IMP in this study. Subjects consented and screened but not dosed in previous phase I studies are not excluded.
18. Current smokers or users of nicotine products. Irregular use of nicotine (e.g. smoking, snuffing, chewing tobacco) less than three times per week is allowed before screening visit.
19. Positive screen for drugs of abuse or alcohol at screening or on admission to the unit prior to administration of the IMP.
20. Current or history of alcohol abuse and/or use of anabolic steroids or drugs of abuse.
21. Intake of xanthine and/or taurine containing energy drinks within two days prior to screening.
22. Plasma donation within one month of screening or blood donation (or corresponding blood loss) during the three months prior to screening.
23. Investigator considers the subject unlikely to comply with study procedures, restrictions and requirements.

    -

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic of CS1 in plasma | up to four weeks
  Plasma concentration of Valproate in plasma

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | up to four weeks
  Adverse event recording in free text

OTHER OUTCOMES:
change in bleeding time | four weeks
  Differences in bleeding time (minutes)
Change in plasma PAI-1 levels | four weeks
  ng/mL
Change in hs-CRP levels | four weeks
  mg/L
Change in platelet numbers | four weeks
  number of platelets per microliter blood
Change in fibrinogen levels | four weeks
  g/L
Change in PAP | four weeks
  ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Bergh, PhD, Study Chair — Cereno Scientific AB
Locations (1):
- CTC Clinical Trial Consultants AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/02/NCT03903302/Prot_SAP_000.pdf